CLINICAL TRIAL: NCT06767800
Title: Phase II Clinical Trial Evaluating the Efficacy and Safety of TQB2102 for Injection in Chemotherapy With Behmosubstituted Monoclonalb/Pembrolizumab ± Chemotherapy in Patients With Unresectable, Locally Advanced, Recurrent, or Metastatic HER2-Positive Gastroesophageal Adenocarcinoma
Brief Title: A Clinical Trial Evaluating TQB2102 for Injection in Combination With Behmosubaisumab/Payamprolizumab With or Without Chemotherapy in Unresectable Locally Advanced, Recurrent, or Metastatic Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Gastroesophageal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2102-II-04
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-08

CONDITIONS: Gastroesophageal Adenocarcinoma
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB2102 for injection (7.5 mg) +Benmelstobart+Chemotherapy (Experimental): TQB2102 for Injection and bemarituzumab are administered intravenously every three weeks, while chemotherapy is given orally from Day 1 to Day 15, with each treatment cycle lasting 21 days.
  TQB2102 and bemosubicinumab for injection every three weeks and capecitabine Day1-Day15 administered orally in 21-day cycles
  Interventions: Drug: TQB2102 for injection (7.5 mg) +Benmelstobart+Chemotherapy
- TQB2102 for injection (6 mg/7.5 mg) +Benmelstobart+Chemotherapy (Experimental): TQB2102 for Injection and bemarituzumab are administered intravenously every three weeks, while chemotherapy is given orally from Day 1 to Day 15, with each treatment cycle lasting 21 days.
  Interventions: Drug: TQB2102 for injection (6 mg/7.5 mg) +Benmelstobart+Chemotherapy
- TQB2102 for injection (6 mg/7.5 mg) +Penpulimab+Chemotherapy (Experimental): TQB2102 for Injection and Penpulimab are administered intravenously every three weeks, while chemotherapy is given orally from Day 1 to Day 15, with each treatment cycle lasting 21 days.
  Interventions: Drug: TQB2102 for injection (6 mg/7.5 mg) +Penpulimab+Chemotherapy

INTERVENTIONS:
Drug: TQB2102 for injection (7.5 mg) +Benmelstobart+Chemotherapy — TQB2102 for injection is an antibody-coupled drug Benmelstobart is a Programmed cell death -Ligand 1 (PD-L1) Antibody
  Arms: TQB2102 for injection (7.5 mg) +Benmelstobart+Chemotherapy
Drug: TQB2102 for injection (6 mg/7.5 mg) +Benmelstobart+Chemotherapy — TQB2102 for injection is an antibody-coupled drug Benmelstobart is a PD-L1 Antibody
  Arms: TQB2102 for injection (6 mg/7.5 mg) +Benmelstobart+Chemotherapy
Drug: TQB2102 for injection (6 mg/7.5 mg) +Penpulimab+Chemotherapy — TQB2102 for injection is an antibody-coupled drug
  Arms: TQB2102 for injection (6 mg/7.5 mg) +Penpulimab+Chemotherapy

SUMMARY:
TQB2102 for injection is a novel antibody-coupled drug (ADC) that enhances binding to tumor cell surface HER2 proteins by simultaneously targeting the two non-overlapping epitopes of the HER2 protein, Endothelial Cell Dysfunction 2 (ECD2) and Endothelial Cell Dysfunction 4 (ECD4), increasing HER2 internalization, and then down-regulating the tumor cell surface HER2 proteins more effectively, and doubly blocking the HER2 signaling, to achieve the effects of trastuzumab and Pertuzumab alone and in combination. This is a Phase II study to evaluate the efficacy and safety of TQB2102 for injection in combination with Benmelstobart Injection /Penpulimab Injection ± chemotherapy in patients with unresectable locally advanced, recurrent or metastatic HER2-positive gastroesophageal adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age, an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, and life expectancy≥3 months;
* Histopathologically confirmed unresectable locally advanced, recurrent or metastatic HER2-positive gastroesophageal adenocarcinoma;
* HER2 expression levels of Immunohistochemistry(IHC) 3+ or IHC 2+ and In Situ Hybridization (ISH) positivity were confirmed in tumor tissue;
* Subject is able to provide previous compliant PD-L1 expression level test results or is able to provide sufficient and competent tumor tissue for PD-L1 expression level testing;
* Patients who have not received prior systemic therapy for locally advanced or metastatic gastric cancer and who have experienced tumor recurrence or metastasis at least 6 months after the completion of prior adjuvant or neoadjuvant therapy may be enrolled;
* Confirmation of at least one measurable lesion according to RECIST 1.1 criteria;
* The main organs function well;
* Male or female patient had no plans to become pregnant and voluntarily take effective contraceptive measures from agree with the study to at least 6 months after the last dose of study drug.

Exclusion Criteria:

* Concurrent secondary malignancy. or other malignancy with no evidence of disease for more than 5 years;
* Uncontrollable toxic reactions above CTC AE grade 1 due to any prior therapy, excluding alopecia;
* Major surgical treatment, incisional biopsy or significant traumatic injury or prolonged unhealed wound or fracture within 28 days prior to first dose;
* Prior history of interstitial lung disease/pneumonia (non-infectious) requiring steroidal drug intervention or current concomitant (or suspected) interstitial lung disease/pneumonia;
* Arterial/venous thrombotic events, such as cerebrovascular accidents, deep vein thrombosis, and pulmonary embolism, have occurred within 6 months prior to the first dose;
* Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;
* Subjects with the presence of any severe and/or uncontrolled disease；
* Subjects who have received other antitumor drugs such as chemotherapy, radiotherapy, or immunotherapy within 4 weeks prior to the first dose, or who are still within the 5 half-life of the drug (whichever occurs shortest); have received a proprietary Chinese medicine with an antitumor indication as specified in the National Medical Products Administration(NMPA) -approved drug insert within 2 weeks prior to the first dose; and have experienced any hemorrhagic or bleeding event in the month prior to the initiation of study treatment ≥CTC Patients with AE grade 3;
* Subjects with known Central nervous system (CNS) metastases and/or carcinomatous meningitis
* Presence of severe bone damage and spinal cord compression due to tumor bone metastases;
* History of live attenuated vaccination within 28 days prior to the first dose or planned live attenuated vaccination during the study;
* History of severe hypersensitivity reactions to large molecule drugs or hypersensitivity to known components of TQB2102, benmelstobart or pembrolizumab for injection;
* Active autoimmune disease requiring systemic therapy (e.g., use of disease-mitigating drugs, corticosteroids, or immunosuppressive agents) within 2 years prior to the first dose of medication
* Diagnosis of immunodeficiency or undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy that was continued within 2 weeks prior to initiation of study treatment.
* Participants who have participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first medication use
* Unstable or serious concurrent medical conditions, as assessed by the Investigators, that would substantially increase the risk-benefit ratio of participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an average of 1 year
  Defined as the percentage of Complete Response (CR) plus partial response (PR) assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria and guidelines for response criteria for use in trials testing immunotherapeutics (iRECIST )for solid tumors.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to disease progression or die, an average of 3 year
  Defined as the time from first use of TQB2102 to first disease progression or death from any cause
Duration of Response (DOR) | Through study completion, an average of 1 year
  Defined as the time from first documented response to documented disease progression or death
Overall survival(OS) | Baseline up to die, an average of 3 year
  Overall survival refers to the time from the first treatment to death from any cause
Number of patients with adverse events (AEs) and serious adverse events (SAEs) | Baseline up to 28 days after the last dose
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (39):
- China (39):
  - Fuyang Cancer Hospital, Fuyang, Anhui
  - Lu'an People's Hospital, Lu'an, Anhui
  - Maanshan People's Hospital, Maanshan, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The first affiliated hospital of chongqing medical university, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Gansu Prouincial Cancer Hospital, Lanzhou, Gansu
  - Gansu Wuwei Tumour Hospital, Wuwei, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - The Second Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The first affiliated hospital of hainan medical university, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The 1st Affiliated Hospital of He'nan University of Science and Technology, Luoyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - NanJing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangning Hospital of Nanjing City, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Fudan university shanghai cancer center, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Nanchong Central Hospital, Nanchong, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Affiliated Cancer Hospital, Ürümqi, Xinjiang
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou, Zhejiang